CLINICAL TRIAL: NCT05555446
Title: In-vivo Study of the Efficacy of Hyperimmune Bovine Colostrum to Block Absorption of Gliadin Peptides in the Human Intestine: a Novel Potential Intervention for Celiac Disease and Non-celiac Gluten Sensitivity
Brief Title: Bovine Colostrum to Prevent Absorption of Gluten
Status: Suspended | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Disengagement from sponsor, no funding provided since 2022.
Sponsor: Milky Way Life Sciences LLC (Industry)
Collaborators: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2019P001133 - clinical
Record Dates: First submitted 2022-09-22; First posted 2022-09-26 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Celiac Disease; Gluten Sensitivity; Non-celiac Gluten Sensitivity
Keywords: celiac disease; gluten; colostrum
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Intervention Model Description: Subjects will subsequently have either the bovine colostrum and then the placebo or vice-versa
Who Masked: Participant, Investigator
Masking Description: Both participant and investigator will not be aware whether subject is having the colostrum or the placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bovine colostrum (Experimental): Participant will receive 18g of bovine colostrum with apple sauce and 1g of gluten.
  Interventions: Dietary Supplement: Bovine colostrum
- Placebo (Placebo Comparator): Participant will receive 18g of placebo with apple sauce and 1g of gluten.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Bovine colostrum — Subject will receive bovine colostrum with gluten.
  Arms: Bovine colostrum
Dietary Supplement: Placebo — Subject will receive a placebo with gluten.
  Arms: Placebo

SUMMARY:
To investigate the use of hyperimmune bovine colostrum to reduce gluten absorption.

A double-blind, cross-over study will be performed in which persons who are following a strict gluten-free diet will be challenged with oral gluten with or without the bovine colostrum.

DETAILED DESCRIPTION:
Physiologic double-blind, cross-over, study in which volunteers on a gluten-free diet will ingest gluten with or without colostrum.

Subject Participation and Study Duration

The study will imply 5 visits for each participant. At the second and fourth visit, they will either take gluten with colostrum powder or with a placebo. Follow-up duration will be until three days after the last study visit.

Each participant will be given daily proton pump inhibitor (PPI) therapy (omeprazole 20 mg) at least one week before the first intervention, and for the entire duration of the study.

Each participant will be invited to fill a celiac disease patient reported outcomes questionnaire (Celiac Disease Symptoms Diary) for the 24 hours prior the study intervention and three days after. Blood and urine samples will be collected during the 24 hours following each study intervention (gluten + colostrum or gluten + placebo)

Adverse events will be recorded during the entire study from enrollment to termination (termination will occur 3 days after the second challenge at the end of the patient reported outcome (PRO) recording period).

ELIGIBILITY:
Inclusion Criteria:

* Self-reported strict adherence to a gluten-free diet for at least 3 months. This may be a lifestyle choice, in solidarity with a child or other family/household member with celiac disease, because of non-celiac gluten sensitivity or because of celiac disease.
* Willing to provide informed consent for all study procedures
* Healthy volunteer according to the investigator assessment (history and physical exam)

Exclusion Criteria:

* Definite or probable gluten exposure during the 72 hours preceding each study intervention visit
* Known active gastrointestinal disease.
* Use of an oral digestive enzyme supplement during the 72 hours preceding each study intervention (challenge) visit.
* History of severe symptomatic reactions to gluten or milk proteins
* History of allergy to beef or meat
* History of allergy to apple
* Severe lactose intolerance
* Any medication or medical condition which, in the opinion of the investigators, could adversely affect the patient's participation in the trial.
* Allergy to PPI or other contraindication for PPI use (i.e history of interstitial nephritis attributed to PPI, history of PPI-induced diarrhea)
* Pregnant women (according to pregnancy test)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-09-22 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Gluten immunogenic peptides in urine | 24 hours
  The main outcome measure will be the intra-subject area under the curve (AUC) for gluten immunogenic peptides measured in urine following gluten challenge with placebo compared to the AUC for gluten immunogenic peptides following gluten challenge combined with colostrum

SECONDARY OUTCOMES:
Symptom score | 24 hours
  Intra-subject maximal CDSD scores within a single domain for the 24 hours following gluten challenge (1-10)

CONTACTS AND LOCATIONS:
Overall Officials: Jocelyn Silvester, MD PhD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No